CLINICAL TRIAL: NCT06775236
Title: A Phase 1b/2 Clinical Study to Evaluate the Safety and Efficacy of SYS6010 as a Monotherapy or in Combination With SYH2051 Compared to Investigator's Choice Chemotherapy in Patients With EGFR-Expressing Advanced Unresectable or Metastatic Solid Tumors, Including But Not Limited to Breast Cancer
Brief Title: Clinical Trial of SYS6010±SYH2051 Versus Chemotherapy in Advanced Breast Cancer and Other Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CSPC Megalith Biopharmaceutical Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYS6010-008
Record Dates: First submitted 2025-01-01; First posted 2025-01-15 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-01

CONDITIONS: Advanced Solid Tumors; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase 1b: Dose escalation and expansion Phase 2: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SYS6010 injection (Experimental): SYS6010 injection 3.2 mg/kg or 3.6 mg/kg, intravenous drip, Q2W
  Interventions: Drug: SYS6010 jnjection
- SYS6010 injection + SYH2051 tablets (Experimental): SYS6010 injection 3.2 mg/kg intravenous drip + SYH2051 60 or 80 mg, oral, Q2W Or SYS6010 injection 3.6 mg/kg intravenous drip + SYH2051 40 or 60 mg, oral, Q2W
  Interventions: Drug: SYS6010 jnjection; Drug: SYH2051 tablets
- Monotherapy Chemotherapy Group (Active Comparator): Investigator's choice of monotherapy chemotherapy （Eribulin, Capecitabine, Gemcitabine, Vinorelbine, or Taxanes. )
  Interventions: Drug: monotherapy chemotherapy

INTERVENTIONS:
Drug: SYS6010 jnjection — SYS6010 is an antibody conjugate drug (ADC), composed of one anti-EGFR monoclonal antibody coupled to one JS1 via an enzyme specific linker
  Arms: SYS6010 injection; SYS6010 injection + SYH2051 tablets
Drug: monotherapy chemotherapy — Investigator's choice of monotherapy chemotherapy (Eribulin, Capecitabine, Gemcitabine, Vinorelbine, or Taxanes.)
  Arms: Monotherapy Chemotherapy Group
Drug: SYH2051 tablets — SYH2051 is a Selective ATM protein kinase inhibitor
  Arms: SYS6010 injection + SYH2051 tablets

SUMMARY:
The study consists of two phases. Phase 1b and Phase 2. Phase 1b aims to evaluate the safety, tolerability, and preliminary efficacy of SYS6010 as a monotherapy and in combination with SYH2051, and to determine the recommended Phase 2 dose (RP2D) for subsequent Phase 2 studies. Phase 2 aims to assess the efficacy and safety of SYS6010 monotherapy or in combination with SYH2051 compared to investigator-selected chemotherapy in patients with EGFR-expressing, unresectable locally advanced or metastatic advanced breast cancer.

DETAILED DESCRIPTION:
Phase Ⅰb Design:

Group A (SYS6010 3.2 mg/kg, Q2W):

Monotherapy Cohort: Planned enrollment of 8-12 breast cancer patients to evaluate the safety and preliminary efficacy of SYS6010 monotherapy.

Combination Cohort: Includes dose-escalation and expansion phases. Dose-escalation phase: A "3+3" design will be used to explore the safety of SYS6010 combined with SYH2051, with SYH2051 doses ranging from 60-80 mg.

Expansion phase: Upon completion of dose-escalation and confirmation of safety, breast cancer patients may be enrolled in the expansion phase.

Group B (SYS6010 3.6 mg/kg, Q2W):

Monotherapy Cohort: Planned enrollment of 8-12 breast cancer patients. Combination Cohort: Similar to Group A, with SYH2051 doses ranging from 40-60 mg.

Group C (SYS6010 3.6 mg/kg, Q2W): Enroll 40 EGFR-expressing HR+/HER2- breast cancer patients to further evaluate the safety and efficacy in this specific population.

Phase Ⅱ Design:

Based on molecular subtypes of breast cancer, cohort studies will be conducted.

Each cohort will enroll 125 patients, randomized in a 2:2:1 ratio into three groups:

SYS6010 + SYH2051 SYS6010 monotherapy Chemotherapy control.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years. 2. Phase 1b/Phase 2: Breast cancer (no tumor type restriction during the combination dose escalation phase).

  3. Provide tumor tissue samples for immunohistochemical EGFR expression testing, with EGFR expression positive as confirmed by the central laboratory.

  4. At least one measurable extracranial lesion according to RECIST v1.1 criteria (no requirement during the combination dose escalation phase of Phase 1b).

  5. ECOG performance status score of 0-1. 6. Expected survival ≥ 3 months. 7. Major organ function meets the relevant laboratory test standards for hematology, renal function, liver function, and coagulation within 7 days prior to treatment.

  8. Subject agrees to use effective contraception from the time of signing the informed consent form until 6 months after the last dose.

  9. Willing to participate in the study, understand the study procedures, and sign a written informed consent form.

Exclusion Criteria:

* 1. Active central nervous system (CNS) metastases or carcinomatous meningitis. Patients with treated and stable brain metastases are eligible for inclusion.

  2. Previously diagnosed HER2-positive breast cancer (IHC 3+ or ISH positive) (Applicable to Phase 1b Group C and Phase 2).

  3. Previously treated with antibody-drug conjugates (ADC) containing topoisomerase I inhibitors (Applicable to Phase 1b Group C and Phase 2).

  4. Allergy to any component of SYS6010 or SYH2051, or to humanized monoclonal antibodies.

  5. Allergy to any component of SYS6010 or SYH2051, or to humanized monoclonal antibodies (This is a repeat of criteria #4).

  6. Adverse events from prior antitumor therapy not recovered to ≤ Grade 1 (unless the investigator deems there is no safety risk).

  7. Failure to meet the required washout period for prior medications or treatments as specified in the protocol.

  8. History of severe cardiovascular or cerebrovascular diseases. 9. History of interstitial lung disease (ILD) / non-infectious pneumonia, or current ILD/non-infectious pneumonia, or imaging findings at screening that cannot rule out these conditions.

  10. Thyroid dysfunction requiring medication, unless the condition is controlled by medication and no dose adjustments are needed.

  11. Severe infection within 4 weeks prior to the first use of the investigational drug.

  12. History of discontinuing EGFR-targeted therapy for ≥ 1 month due to skin toxicity, or current skin conditions requiring medication.

  13. Gastrointestinal diseases or functional impairments that may significantly affect the absorption of the investigational drug (e.g., ulcerative disease, severe nausea/vomiting, diarrhea, malabsorption, etc.).

  14. Uncontrolled pleural or peritoneal effusion. 15. Active HBV or HCV infection, syphilis, HIV infection, or AIDS. 16. Other conditions deemed by the investigator as unsuitable for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity(DLT) occurrence and incidence | Up to approximately 3 months after the first participant is enrolled
  The occurrence and incidence of dose-limiting toxicities (DLTs) will be assessed based on predefined criteria during the first 28 days after the initial dose. DLTs are defined as adverse events related to the study drug that meet the protocol-specified criteria for dose limitation.
Adverse events (AE) occurrence and incidence | Up to approximately 36 months after the first participant is enrolled
  The occurrence and incidence of adverse events (AEs) will be evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. AEs will be monitored from the first dose until the safety follow-up period.
Objective response rate (ORR) per RECIST v1.1 | Up to approximately 36 months after the first participant is enrolled
  The objective response rate (ORR) will be assessed based on RECIST v1.1 criteria. ORR is defined as the proportion of patients achieving a complete response (CR) or partial response (PR) as the best overall response.

SECONDARY OUTCOMES:
Disease control rate (DCR) per RECIST 1.1 | Up to approximately 36 months after the first participant is enrolled
Duration of response (DoR) per RECIST 1.1 | Up to approximately 36 months after the first participant is enrolled
Progression free survival (PFS) per RECIST 1.1 | Up to approximately 36 months after the first participant is enrolled
Overall survival(OS) | Up to approximately 36 months after the first participant is enrolled
PK parameters of toxin-bound antibody | Up to approximately 36 months after the first participant is enrolled
Description :total antibody and free toxin (JS-1) after single and continuous administration of SYS6010 | Up to approximately 36 months after the first participant is enrolled
PK parameters after single and multiple administrations of SYH2051 | Up to approximately 36 months after the first participant is enrolled